CLINICAL TRIAL: NCT05754086
Title: A Multidimensional Study on Articulation Deficits in Parkinson's Disease
Brief Title: A Multidimensional Study on Articulation Deficits in Parkinsons Disease
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Yunjung Kim, Principal Investigator, Florida State University
Other Study IDs: STUDY00002525; F31DC020121 (NIH)
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease; Dysarthria, Hypokinetic
MeSH Terms: conditions — Parkinson Disease; Dysarthria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinsons (PD) Group: This cohort includes individuals who have been diagnosed with Parkinson's disease.
  Interventions: Behavioral: Clear Speech; Behavioral: Less Clear Speech
- Neurotypical (NT) Group: This group consists of age-matched control participants. They are neurologically healthy and do not have any neurological diagnoses.
  Interventions: Behavioral: Clear Speech; Behavioral: Less Clear Speech

INTERVENTIONS:
Behavioral: Clear Speech — This behavioral modification asks participants to speak more clearly, as if they were "speaking to someone with a hearing loss".
Behavioral: Less Clear Speech — This behavioral modification asks participants to speak less clearly, as if they were "in a room with many people and they were mumbling something to the person next to them that they didn't want other people in the room to hear."

SUMMARY:
Articulatory deficits are present in most speakers with dysarthria, which negatively impacts their speech intelligibility, yet little is known about the relationship between articulatory movement and speech intelligibility. This study will examine the relationship between articulation measures, both acoustic and kinematic, and their relationship to perceptual measures (i.e., speech intelligibility and articulation ratings) in 30 individuals with dysarthria secondary to Parkinson's disease and 30 neurologically healthy adults of the same age. The findings will have implications for behavioral management.

DETAILED DESCRIPTION:
Dysarthria is a motor speech disorder that affects individuals with various etiologies. Parkinson's disease (PD) alone affects nearly one million individuals in the U.S., with dysarthria developing in approximately 90% of these individuals within the first two years of onset. The dysarthria associated with PD is characterized by reduced movement, which has been supported by findings of reduced lip, tongue, and jaw movement in speakers with PD. However, it remains unclear if hypokinetic dysarthria causes a global reduction across all articulators, or if specific articulators are disproportionally affected by the disease. Further, it is not fully understood what factors contribute to speech intelligibility. Specifically, little is known about the articulatory-kinematic correlates of speech intelligibility. This missing link is vital to understand, as articulation deficits are a universal characteristic of dysarthria, regardless of etiology. The proposed study provides a linked investigation of kinematic, acoustic, and perceptual characteristics in speakers with PD and neurologically healthy speakers.

This research aims to (1) examine the perceptual, acoustic, and articulator-specific movement deficits in speakers with PD and (2) understand the relationship between articulatory movement and measures of speech perception. Specific Aim 1 will examine the group differences between speakers with PD and neurologically healthy speakers using perceptual, acoustic, and articulator-specific kinematic measures. The investigators hypothesize the perceptual, acoustic, and tongue-related kinematic measures will differentiate individuals with PD from neurologically healthy speakers. Specific Aim 2 will model speech intelligibility (Specific Aim 2a) and ratings of articulatory precision (Specific Aim 2b) using selected acoustic and kinematic measurements. The investigators hypothesize that the acoustic measures will be stronger predictors of speech intelligibility than the kinematic measures, as they are both derived from the speech signal. Further, the investigators hypothesize the selected kinematic measures may demonstrate a stronger relationship to articulation ratings than speech intelligibility. This study is a requisite step toward our long-term goal of advancing dysarthria management strategies. The primary outcome will be explanatory models that identify acoustic and articulatory correlates of speech intelligibility and articulatory precision. This study has important implications for developing articulator-specific dysarthria management strategies to supplement universal dysarthria management strategies.

ELIGIBILITY:
Inclusion Criteria:

* neurological diagnosis of PD (for the PD group only)
* diagnosis of dysarthria (for the PD group only)
* native English speaker
* no evidence of cognitive impairment, as indicated by a score above 26 on the Montreal Cognitive Assessment
* able to read a paragraph in 19-point font

Exclusion Criteria:

* Not within the age limits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited via convenient sampling from Tallahassee, FL, and the local community. For the neurologically healthy control speakers, flyers will be posted at local coffee shops, community samples, and via word of mouth. For the Parkinson's participants, flyers will be posted at hospitals, health clinics, and gyms.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Vowel Space Area | Baseline
  Vowel space area is a measure of the planar area among the four corner vowels /i/, /ae/, /a/, and /u/. It is calculated using the first and second formant resonant frequencies obtained from the acoustic signal, using the software PRAAT.
F2 Slope | Baseline
  Second formant frequency (F2) slope is measured as the rate of F2 change during the diphthong in "Buy." To calculate this measure, first the investigators will obtain the extent of F2 change (max F2 - min F2) from the diphthong "Buy." Then this F2 change is divided by the duration of the diphthong "Buy."
Tongue and Jaw Speed | Baseline
  This is measured as the tongue and jaw speed during the diphthong in "Buy". Specifically, this will be calculated as tongue/jaw movement (measured in mm), divided by movement duration (measured in ms). The tongue and jaw movement will be collected using the electromagnetic articulography (EMA) device used in this study.
Acoustic Distance | Baseline
  This is measured as the Euclidean distance between the second formant frequency (F2) onset and offset of the diphthong in "Buy" in an F1-F2 (first and second formant frequency) space. Measured in Hz.
Tongue and Jaw Distance | Baseline
  This is measured as the Euclidean distance between the tongue and jaw onset and offset of the diphthong in "Buy" in a two-dimensional space.The tongue and jaw movement will be collected using the electromagnetic articulography (EMA) device used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Yunjung Kim, Ph.D., Study Chair — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The analytic data and code will be shared to the open science framework (OSF) upon completion of the project, expected July 2023.
Supporting Information: Analytic Code
Time Frame: Analytic data and code will be made available in July 2023.
Access Criteria: Upon publication to the open science framework (OSF) project page, anyone will have access to the analytic data and code.
URL: https://osf.io/hfuq5/

DOCUMENTS (1):
  • Informed Consent Form (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT05754086/ICF_000.pdf